CLINICAL TRIAL: NCT02069392
Title: Nicotinic Enhancement of Cognitive Remediation Training in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Britta Hahn, Associate Professor (Britta Hahn, Ph.D.), University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00058233; R21MH095824 (NIH)
Record Dates: First submitted 2014-02-05; First posted 2014-02-24 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; cognition; cognitive remediation; nicotine
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — halofantrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive remediation training with nicotine (Active Comparator): Participants will complete daily sessions of Posit Science cognitive remediation training for 10 weeks. Twice a week, participants will consume a 2 mg (for non-smokers) or 4 mg (for smokers) nicotine polacrilex lozenge prior to the training.
  Interventions: Behavioral: Cognitive remediation training; Drug: Nicotine polacrilex lozenge
- Cognitive remediation training without nicotine (Placebo Comparator): Participants will complete daily Posit Science cognitive remediation training for 10 weeks. Twice a week, participants will consume a placebo lozenge prior to the training.
  Interventions: Behavioral: Cognitive remediation training

INTERVENTIONS:
Behavioral: Cognitive remediation training
  Other Names: Posit Science cognitive remediation training
Drug: Nicotine polacrilex lozenge — Of interest are the effects of nicotine on cognitive remediation training benefits.
  Other Names: Nicorette polacrilex lozenges, GlaxoSmithKline, 2 mg and 4 mg
  Arms: Cognitive remediation training with nicotine

SUMMARY:
Schizophrenia is marked by problems in attention, memory and problem solving. These deficits predict long-term functional outcome such as the ability to live independently and maintain employment, but they are not ameliorated by currently available medications. Cognitive training improves these functions to some degree, but this approach is time- and resource-intensive. The current project aims at enhancing and accelerating the benefits that people with schizophrenia derive from cognitive training by administering nicotine during some of the training sessions. This would provide the proof of principle for a type of treatment intervention to improve cognitive symptoms of schizophrenia.

The current project aims at determining whether the intermittent presence of nicotine during cognitive training exercises in people with schizophrenia will shorten the training period necessary to induce significant and clinically relevant improvement and enhance the improvement seen after a training period of specified length.

Hypothesis 1a: Nicotine administration during training will increase the size of all measured effects of the training intervention, and will accelerate the time course of performance enhancement on the MCCB and training exercise progression parameters.

Hypothesis 1b: The larger training effects in the Nicotine Group will persist beyond the end of the intervention.

Hypothesis 2a: Within-session progress on the training exercises will be larger in the presence of nicotine than in the presence of placebo.

Hypothesis 2b: These acute nicotine-induced performance elevations will persist beyond the presence of nicotine through subsequent non-drug training sessions, giving evidence of an acute facilitation of learning processes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60 years.
* DSM diagnosis of schizophrenia or schizoaffective disorder.
* Ability to give written informed consent.
* Either currently smoking and not attempting to quit, or having smoked no more than 80 cigarettes, cigarillos or cigars in lifetime and not at all within the last year.
* Normal or corrected to normal vision (at least 20/50).
* Four weeks of stable pharmacological treatment (same psychiatric medication at same dose) and no foreseeable changes at enrollment.

Exclusion Criteria:

* Alcohol or substance abuse or dependence other than nicotine within the last 12 months.
* Uncontrolled hypertension (resting systolic blood pressure above 150 or diastolic above 90 mm Hg).
* History of myocardial infarction, heart failure, angina, stroke or severe arrhythmias.
* ECG abnormalities.
* History of neurological conditions such as stroke, seizures, dementia or organic brain syndrome.
* Mental retardation.
* Pregnant, verified by urine pregnancy test for females.
* Breast-feeding.
* Treated with benztropine currently or within the last four weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2015-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Britta Hahn, Ph.D., Principal Investigator — University of Maryland School of Medicine, Maryland Psychiatric Research Center
Locations (1):
- Maryland Psychiatric Research Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Remediation Training With Nicotine: Participants complete daily sessions of Posit Science cognitive remediation training for 10 weeks. Twice a week, participants consume a 2 mg (for non-smokers) or 4 mg (for smokers) nicotine polacrilex lozenge prior to the training.
  Cognitive remediation training
  Nicotine polacrilex lozenge: Of interest are the effects of nicotine on cognitive remediation training benefits.
- Cognitive Remediation Training Without Nicotine: Participants complete daily Posit Science cognitive remediation training for 10 weeks. Twice a week, participants consume a placebo lozenge prior to the training.
  Cognitive remediation training
Period: Overall Study
Arm/Group | Cognitive Remediation Training With Nicotine | Cognitive Remediation Training Without Nicotine
Started | 14 | 17
Completed | 10 | 15
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Remediation Training With Nicotine | Cognitive Remediation Training Without Nicotine | Total
Number analyzed (Participants) | 14 | 17 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 17 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (11.0) | 43.8 (12.0) | 43.5 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 10 | 13 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 13 | 17 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 7 | 9 | 16
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 17 | 31
Smoking status [Count of Participants; unit: Participants]
  Smokers | 6 | 7 | 13
  Non-smoker | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: MATRICS Consensus Cognitive Battery (MCCB) Composite Score
Description: The MCCB is an FDA-approved assessment tool for trials of cognition-enhancing treatments in people with schizophrenia. The MCCB is comprised of the following domains: 1) Speed of Processing; 2) Attention/Vigilance; 3) Working Memory; 4) Verbal Learning; 5) Visual Learning; 6) Reasoning and Problem Solving; and 7) Social Cognition. The composite score is standardized to a T-scale (mean=50, standard deviation=10) based on healthy control normative data. Better performance is reflected by higher scores.
Time Frame: baseline (week 0), weeks 4 and 7 of intervention, end-of-intervention (week 10), 4-week follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Remediation Training With Nicotine | Cognitive Remediation Training Without Nicotine
Number analyzed (Participants) | 10 | 15
score on a scale
  Baseline | 32.30 (15.42) | 33.87 (10.40)
  Week 4 | 32.50 (14.98) | 35.47 (9.02)
  Week 7 | 35.30 (13.70) | 36.87 (9.75)
  Week 10 (end of intervention) | 34.60 (14.38) | 36.67 (10.27)
  4-week follow-up | 35.00 (12.67) | 37.87 (10.14)

2. Secondary Outcome: Cognitive Assessment Interview (CAI) Score
Description: Clinician-administered interview about daily life cognitive functioning. The CAI assesses 10 items related to working memory, attention/vigilance, learning/memory, problem solving, processing speed, and social cognition. The total score ranges from 1 (inability to maintain personal hygiene due to cognitive deficits) to 100 (superior cognitive functioning in a wide range of activities). A score of 55 corresponds to moderate cognitive symptoms, e.g. persistent problems paying attention or forgetting scheduled events.
Time Frame: baseline (week 0) and post-intervention (week 10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Remediation Training With Nicotine | Cognitive Remediation Training Without Nicotine
Number analyzed (Participants) | 10 | 15
score on a scale
  Baseline | 55.80 (12.88) | 59.14 (9.59)
  Post-intervention (week 10) | 69.30 (12.52) | 64.79 (10.69)

3. Secondary Outcome: Change in Abbreviated Schizophrenia Quality of Life Scale Score
Description: Semi-structured clinician interview measuring functional outcome and quality of life in people with schizophrenia. Includes subjective questions regarding life satisfaction and objective indicators of social and occupational role functioning during preceding 4 weeks. Seven items are scored on a 0 (severe impairment) to 6 (high functioning) scale. The total score ranges from 0 to 42, with larger values reflecting higher functioning.
Time Frame: baseline (week 0) and post-intervention (week 10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Remediation Training With Nicotine | Cognitive Remediation Training Without Nicotine
Number analyzed (Participants) | 10 | 15
score on a scale
  Baseline | 22.30 (5.70) | 20.29 (5.99)
  Post-intervention (week 10) | 24.90 (5.88) | 23.00 (4.02)

4. Secondary Outcome: UCSD Performance-Based Skills Assessment (UPSA) Score
Description: Measures ability to perform real-life tasks by standardized role-play. Scores reflect percent correct, i.e. range from 0-100 with higher scores representing better performance.
Time Frame: baseline (week 0) and post-intervention (week 10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Remediation Training With Nicotine | Cognitive Remediation Training Without Nicotine
Number analyzed (Participants) | 10 | 15
score on a scale
  Baseline | 77.50 (14.97) | 71.87 (14.01)
  Post-intervention (week 10_ | 75.50 (14.55) | 74.00 (12.28)

5. Secondary Outcome: Calgary Depression Scale Score
Description: Clinician scale developed to assess the level of depression in schizophrenia. 9 items assess symptoms of depression and overall rater impression on a scale from 0 (absent) to 3 (severe).
Time Frame: baseline (week 0), post-intervention (week 10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Remediation Training With Nicotine | Cognitive Remediation Training Without Nicotine
Number analyzed (Participants) | 10 | 15
score on a scale
  Baseline | 2.40 (2.45) | 2.07 (2.28)
  Post-intervention (10 weeks) | 2.50 (2.59) | 1.40 (1.59)

6. Secondary Outcome: Scale for the Assessment of Negative Symptoms (SANS) Score
Description: Clinician rating scale of negative symptoms in schizophrenia. Within each of 5 domains, separate symptoms are rated from 0 (absent) to 5 (severe). Total scores are the sum of 22 subscales and range from 0 to 110, with larger values reflecting higher negative symptoms.
Time Frame: baseline (week 0), post-intervention (week 10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Remediation Training With Nicotine | Cognitive Remediation Training Without Nicotine
Number analyzed (Participants) | 10 | 15
score on a scale
  Baseline | 36.40 (11.64) | 37.73 (7.09)
  Post-intervention (10 weeks) | 33.80 (12.14) | 36.53 (7.04)

7. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS) Score
Description: Clinician rating scale to measure psychotic symptoms. Each of 20 items is scored 1-7. Total scores are the sum of all items and range from 20 to 140, with larger values reflecting worse symptoms.
Time Frame: baseline (week 0), post-intervention (week 10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Remediation Training With Nicotine | Cognitive Remediation Training Without Nicotine
Number analyzed (Participants) | 10 | 15
score on a scale
  Baseline | 39.40 (9.14) | 37.33 (7.87)
  Post-intervention (10 weeks) | 39.50 (9.43) | 36.53 (5.55)

8. Secondary Outcome: Training Exercise Parameters: Visual and Sound Sweeps
Description: Some of the Posit Science exercises provide an assessment tool of training progress on task parameters, which adjust continuously to keep performance at ~85% correct. Enhanced sensory processing speed and precision is considered the central building block of training benefits. Therefore, we analyzed the two exercises aimed at training these processes. Performance is quantified as stimulus presentation time in ms of visual or sound "sweeps", which the participant has to judge in terms of change across space or time. Smaller values reflect better performance. Visual and sound sweeps were averaged.
Time Frame: baseline (week 0), post-intervention (week 10), 4-week follow-up
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Cognitive Remediation Training With Nicotine: Participants will complete daily sessions of Posit Science cognitive remediation training for 10 weeks. Twice a week, participants will consume a 2 mg (for non-smokers) or 4 mg (for smokers) nicotine polacrilex lozenge prior to the training.
  Cognitive remediation training
  Nicotine polacrilex lozenge: Of interest are the effects of nicotine on cognitive remediation training benefits.
- Cognitive Remediation Training Without Nicotine: Participants will complete daily Posit Science cognitive remediation training for 10 weeks. Twice a week, participants will consume a placebo lozenge prior to the training.
  Cognitive remediation training
Arm/Group | Cognitive Remediation Training With Nicotine | Cognitive Remediation Training Without Nicotine
Number analyzed (Participants) | 10 | 15
ms
  Baseline | 130.25 (46.26) | 198.80 (159.16)
  Week 10 (end-of-treatment) | 94.40 (28.04) | 124.40 (73.03)
  4-week follow-up | 102.80 (39.45) | 117.50 (69.76)

9. Secondary Outcome: Change in Working Memory Capacity
Description: Derived from a computerized change localization task. One to four colored squares are shown for 100 ms. After a delay, they reappear and the task is to click on the one square that has changed color (50% chance). Performance is expressed as the percentage of correct responses.
Time Frame: baseline (week 1) and post-intervention (week 10)
Measure: Mean (Standard Deviation); unit: percentage correct responses
Arm/Group | Cognitive Remediation Training With Nicotine | Cognitive Remediation Training Without Nicotine
Number analyzed (Participants) | 10 | 15
percentage correct responses
  Baseline | 67.7 (16.0) | 67.5 (14.5)
  Post-intervention (10 weeks) | 67.2 (13.7) | 68.6 (13.7)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 10 weeks of exposure to cognitive remediation training with bi-weekly exposure to nicotine or placebo.
Arm/Group | Cognitive Remediation Training With Nicotine | Cognitive Remediation Training Without Nicotine
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/17
Other Adverse Events (participants affected / at risk) | 0/14 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT02069392/Prot_SAP_000.pdf